CLINICAL TRIAL: NCT04573426
Title: Effects of Acetaminophen on Pain Response Among Overweight or Obese Women Exposed to Weight Stigmatization
Brief Title: Pain and Acetaminophen in Women Study
Acronym: PAWS
Status: Completed | Type: Observational
Sponsor: Ohio State University (Other)
Responsible Party: Principal Investigator, Charles Emery PhD, Professor of Psychology, Ohio State University
Other Study IDs: 2019H0381
Record Dates: First submitted 2020-09-14; First posted 2020-10-05 (Actual); Last update posted 2021-09-08 (Actual); Status verified 2021-09

CONDITIONS: Overweight; Obesity; Healthy Adults
Keywords: Weight stigma; Stigma; Overweight; Obesity; Acetaminophen; Inflammation; Analgesics; Anti-inflammatory
MeSH Terms: conditions — Overweight; Obesity; Weight Prejudice; Social Stigma; Inflammation | interventions — Acetaminophen

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Saliva and dried blood spots (both frozen after collection)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

GROUPS / COHORTS (5):
- Overweight/Obese+Drug+Stigma: 40 participants with overweight or obesity will consume 1,000mg of acetaminophen in a liquid vehicle briefly following the start of the appointment. After one hour, they will read a short vignette meant to induce weight stigma.
  Interventions: Drug: Acetaminophen; Behavioral: Weight stigma vignette
- Overweight/Obese+Drug+Control: 40 participants with overweight or obesity will consume 1,000mg of acetaminophen in a liquid vehicle briefly following the start of the appointment. After one hour, they will read a short control vignette meant to have no impact on their emotional state.
  Interventions: Drug: Acetaminophen; Behavioral: Control vignette
- Overweight/Obese+Placebo+Stigma: 40 participants with overweight or obesity will consume a placebo solution briefly following the start of the appointment. After one hour, they will read a short vignette meant to induce weight stigma.
  Interventions: Drug: Placebo; Behavioral: Weight stigma vignette
- Overweight/Obese+Placebo+Control: 40 participants with overweight or obesity will consume a placebo solution briefly following the start of the appointment. After one hour, they will read a short control vignette meant to have no impact on their emotional state.
  Interventions: Drug: Placebo; Behavioral: Control vignette
- Normal Weight+Placebo+Stigma: 40 participants with normal weight will consume a placebo solution briefly following the start of the appointment. After one hour, they will read a short vignette meant to induce weight stigma.
  Interventions: Drug: Placebo; Behavioral: Weight stigma vignette

INTERVENTIONS:
Drug: Acetaminophen — 1,000mg liquid acetaminophen
  Groups: Overweight/Obese+Drug+Control; Overweight/Obese+Drug+Stigma
Drug: Placebo — Liquid placebo solution
  Groups: Normal Weight+Placebo+Stigma; Overweight/Obese+Placebo+Control; Overweight/Obese+Placebo+Stigma
Behavioral: Weight stigma vignette — Short vignette meant to induce weight stigma by describing one's rejection for a promotion due to their weight
  Groups: Normal Weight+Placebo+Stigma; Overweight/Obese+Drug+Stigma; Overweight/Obese+Placebo+Stigma
Behavioral: Control vignette — Short vignette meant to have no effect on emotion describing a generic promotion process
  Groups: Overweight/Obese+Drug+Control; Overweight/Obese+Placebo+Control

SUMMARY:
The purpose of this study is to evaluate the influence of acetaminophen on pain response and inflammation.

DETAILED DESCRIPTION:
The purpose of this study is to evaluate the influence of weight stigma on emotional functioning and biomarkers of inflammation among overweight and obese women; and to determine the degree to which acetaminophen moderates the stigma-related effects. Participants will provide blood spot and saliva samples upon arrival, and then be randomly assigned to consume either 1,000mg of acetaminophen in liquid form, or a placebo solution. Participants then will complete a series of questionnaires assessing a variety of relevant psychological and behavioral constructs. After this participants will be randomly assigned to read one of two shorts stories and answer a series of questions about their reaction to the story. Finally, participants will answer another series of questionnaires and provide a second saliva sample. Participants will first be adult women in the Columbus, Ohio and surrounding areas with body mass indices considered overweight or obese. A smaller cohort of women with normal weight will be recruited at a later time for purposes of comparison.

ELIGIBILITY:
Inclusion Criteria:

* At least 18 years old and biologically female

Exclusion Criteria:

* Due to the use of acetaminophen in this study, women who report current pregnancy will be excluded from the study due to potential negative effects on pregnancy.

The following are additional exclusion criteria:

1. Visual impairment that would impair one's ability to read to the extent that they could not read items on paper or a computer screen.
2. Stopping schooling prior to completing ninth grade.
3. A history of liver disorder and/or alcohol abuse.
4. A current prescription of a drug that contains acetaminophen.
5. Allergy to acetaminophen
6. A score on the Patient Health Questionnaire - 9 depressive symptom scale of 15 or greater.
7. For normal weight participants, a history of overweight or obesity.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: 160 women with overweight or obesity from the Columbus, Ohio and surrounding areas who also meet other study criteria will be recruited for the study. A smaller cohort of 40 women with normal weight who meet the same study criteria, and deny a history of overweight or obesity, will also be recruited. All participants will be 18 years of age or older
Sampling Method: Non-Probability Sample
Enrollment: 200 (Actual)
Dates: Start 2019-11-15 (Actual); Primary Completion 2021-05-02 (Actual); Study Completion 2021-05-02 (Actual)

PRIMARY OUTCOMES:
Baseline Prostaglandin level | Within the first 10 minutes of the two-hour session
  Prostaglandin level (measured via PGE2) will be assessed via saliva and will be utilized as an objective marker of baseline inflammation Baseline prostaglandin level will be determined by analyzing saliva collected within the first ten minutes of the single, two-hour session.
Change in Prostaglandin level | Within the first 10 minutes of the two-hour session and approximately ten minutes prior to the end of the two-hour session.
  Change in prostaglandin level (measured via PGE2) will be assessed via difference in two saliva samples and will be utilized as an objective marker of change in inflammation over the course of the two-hour session. Change in prostaglandin level will be determined by calculating the difference between PGE2 level within the first 10 minutes of the two-hour session, and level of prostaglandins via saliva collection approximately ten minutes prior to ending the two-hour session.
Baseline C-Reactive Protein | Within the first 10 minutes of the two-hour session.
  C-Reactive Protein (CRP) will be determined via dried blood spot analysis. The dried blood spots are collected within the first 10 minutes of the single, two-hour session. This CRP will be used an as objective measure of baseline inflammation.
McGill Pain Questionnaire (baseline) | In the first hour of the two-hour session.
  The McGill Pain Questionnaire (MPQ) will be used to assess baseline pain severity across sensory, affective, evaluative, and miscellaneous qualities of pain. Pain severity scores may range from 0-78 with high scores reflecting greater pain severity. The MPQ also consists of an overall pain intensity scale ranging from 0-5, with higher scores reflecting greater present pain intensity. Baseline pain will be measured via an MPQ administered with a set of questionnaires in the first hour of the two-hour session.
McGill Pain Questionnaire (change) | Within the first hour and again within the final 30 minutes of the two-hour session.
  The McGill Pain Questionnaire (MPQ) will also be used to assess change in pain severity across sensory, affective, evaluative, and miscellaneous qualities of pain. Pain severity scores may range from 0-78 with high scores reflecting greater pain severity. The MPQ also consists of an overall pain intensity scale ranging from 0-5, with higher scores reflecting greater present pain intensity. Change in pain will be measured by calculating the difference in MPQ score at baseline and the score from the second MPQ administration, which is administered within the final 30 minutes of the two-hour session.
Visual Analog Scale for Pain (baseline) | In the first hour of the two-hour session.
  The Visual Analog Scale for Pain (VAS-Pain) will also be used to measure pain. This is a unidimensional measure of physical pain intensity consisting of a line measuring 100 millimeters anchored by two descriptors representing the extremes of pain: "no pain" versus "my pain is as bad as it could possibly be." Participants mark on the line to indicate their current level of pain. Scores range from 0-100 with higher scores, or greater pain intensity, represented by mark's made farther from the "no pain" anchor. Baseline pain will be measured via a VAS-Pain administered with a set of questionnaires in the first hour of the two-hour session.
Visual Analog Scale for Pain (change) | Within the first hour and again within the final 30 minutes of the two-hour session.
  The Visual Analog Scale for Pain (VAS-Pain) will also be used to measure pain. This is a unidimensional measure of physical pain intensity consisting of a line measuring 100 millimeters anchored by two descriptors representing the extremes of pain: "no pain" versus "my pain is as bad as it could possibly be." Participants mark on the line to indicate their current level of pain. Scores range from 0-100 with higher scores, or greater pain intensity, represented by mark's made farther from the "no pain" anchor. Change in pain will be measured by calculating the difference in VAS-Pain score at baseline and the score from the second VAS-Pain administration, which is administered within the final 30 minutes of the two-hour session.
Stigma Situations Inventory | In the first hour of the two-hour session.
  The Stigma Situations Inventory (SSI) is a 50-item questionnaire of lifetime frequency of obesity-related experiences rated on a 0 (never) to 9 (daily) scale. A higher mean score across all items suggesting greater experience of weight stigma. SSI is administered with a series of questionnaires in the first hour of the two-hour session and will provide a baseline measure of weight stigma experience.
Weight Bias Internalization Scale | In the first hour of the two-hour session.
  The Weight Bias Internalization Scale (WBIS) is an 11-item scale measuring individuals' belief that anti-fat attitudes are relevant to the self. Items are answered on a 7-point Likert scale ranging from 1 (strongly disagree) to 7 (strongly agree), with total scores ranging from 11 to 77. WBIS is administered with a series of questionnaires in the first hour of the two-hour session and will provide a baseline measure of belief that anti-fat attitudes are relevant to the self.
Stigma Impact Scale | In the first hour of the two-hour session.
  The Stigma Impact Scale (SIS) is a 24-item measure used to evaluate the impact of perceived stigma among those with chronic illnesses. The term 'illness' has been changed to 'condition' to enhance applicability to participants in this study. Each item is rated on a 5-point Likert scale ranging from 0 (not applicable) to 4 (strongly agree). Total scores range from 0-96, with higher scores reflecting greater perceived impact of stigma. SIS is administered with a series of questionnaires in the first hour of the two-hour session and will provide a baseline measure of perceived impact of condition, in this case obesity, on the respondent.
Impact of Weight on Quality of Life | In the first hour of the two-hour session.
  The Impact of Weight on Quality of Life-Lite (IWQOL-Lite) is a 31-item measure of obesity-related quality of life. Each item is rated on a 5-point Likert scale. Total scores range from 31 to 155 with higher scores reflecting greater impact of weight on quality of life. IWQOL-Lite is administered with a series of questionnaires in the first hour of the two-hour session and will provide a baseline measure of impact of weight on quality of life.
Medical Outcomes Survey, Short-Form-36 | In the first hour of the two-hour session
  The Medical Outcomes Survey, Short Form-36 (SF-36) is a 36-item measure of health-related quality of life. Mental and physical quality of life scores are calculated into a 0-100 scale, with higher scores reflecting better health-related quality of life. SF-36 is administered with a series of questionnaires in the first hour of the two-hour session and will provide a baseline measure of health-related quality of life.
Positive and Negative Affect Schedule (baseline) | In the first hour of the two-hour session
  The Positive and Negative Affect Schedule (PANAS) is a 20-item measure of positive and negative affect. A 5-point Likert scale is used to indicate the degree to which one is experiencing an emotion during the present moment. Total scores for the negative and positive affect subscales range from 10-50. PANAS is administered with a series of questionnaires in the first hour of the two-hour session and will provide a baseline measure of present moment emotional experience.
Positive and Negative Affect Schedule (change) | Within the first hour and again within the final 30 minutes of the two-hour session.
  The Positive and Negative Affect Schedule (PANAS) is a 20-item measure of positive and negative affect. A 5-point Likert scale is used to indicate the degree to which one is experiencing an emotion during the present moment. Total scores for the negative and positive affect subscales range from 10-50. Change in PANAS will be calculated and represent a change in present moment emotional experience during the course of the session. This will be calculated by determining the difference between PANAS scores at baseline and the second PANAS administration, which is administered within the final 30 minutes of the two-hour session.
Visual Analog Scale for Distress (baseline) | In the first hour of the two-hour session
  The Visual Analog Scale for Distress (VAS-Distress) is a unidimensional measure of distress intensity consisting of a line measuring 100 millimeters anchored by two descriptors representing the extremes of distress: "no distress" versus "as distressed as I could possibly be." Participants mark on the line to indicate their current level of distress. Scores range from 0-100 with higher scores, or greater distress intensity, represented by mark's made farther from the "no distress" anchor. Baseline distress will be measured via a VAS-Distress administered with a set of questionnaires in the first hour of the two-hour session.
Visual Analog Scale for Distress (change) | Within the first hour and again within the final 30 minutes of the two-hour session.
  The Visual Analog Scale for Distress (VAS-Distress) is a unidimensional measure of distress intensity consisting of a line measuring 100 millimeters anchored by two descriptors representing the extremes of distress: "no distress" versus "as distressed as I could possibly be." Participants mark on the line to indicate their current level of distress. Scores range from 0-100 with higher scores, or greater distress intensity, represented by mark's made farther from the "no distress" anchor. Change in distress will be measured by calculating the difference in VAS-Distress score at baseline and the score from the second VAS-Distress administration, which is administered within the final 30 minutes of the two-hour session.

SECONDARY OUTCOMES:
International Physical Activity Questionnaire - Short Form | In the first hour of the two-hour session
  The International Physical Activity Questionnaire - Short Form (IPAQ-SF) measures physical activity and inactivity performed during the previous seven days. Respondents report the number of days, hours per day, and minutes per day in the last seven days they engaged in vigorous exercise, moderate exercise, walking, and sitting. The IPAQ-SF will be administered with a set of questionnaires in the first hour of the two-hour session.
Pittsburgh Sleep Quality Index | In the first hour of the two-hour session
  The Pittsburgh Sleep Quality Index (PSQI) is used to assess sleep behavioral (quality and disturbances) over a one-month interval. The PSQI yields a total score (ranging 0-21) as well as the following seven subscales (ranging 0-3): subjective sleep quality, sleep latency, sleep duration, habitual sleep efficiency, sleep disturbances, use of sleep medications, and daytime dysfunction. Higher scores reflect worse sleep quality. The PSQI will be administered with a set of questionnaires in the first hour of the two-hour session.
Rosenberg Self-Esteem Scale | In the first hour of the two-hour session
  The Rosenberg Self-Esteem Scale (RSES) is a 10-item measure used to assess overall self-esteem. Both positive and negative feelings about the self are measured. Items are answered on a Likert scale ranging from 0 (strongly agree) to 3 (strongly disagree), with higher scores indicating higher self-esteem. The RSES will be administered with a set of questionnaires in the first hour of the two-hour session.
Need Threat Scale | In the first hour of the two-hour session
  The Need Threat Scale is a 12-item measure designed to assess one's need for belonging, self-esteem, control, and meaningful existence, each of which represent a subscale of the measure. Respondents indicate how they are feeling right now using a five-point Likert scale ranging from "not at all" to "very much so." In addition to four subscale scores, a composite score is calculated by averaging responses across the 12 items, with lower scores reflecting less needs satisfaction (i.e., more need threat). The Need Threat Scale will be administered with a set of questionnaires in the first hour of the two-hour session.
Hospital Anxiety and Depression Scale | In the first hour of the two-hour session
  The Hospital Anxiety and Depression Scale (HADS) is a 14-item measure developed to assess depression and anxiety among non-psychiatric medical patients. Respondents are asked to rate each item on a scale ranging from 0 (not at all) to 3 (most of the time). The HADS consists of a total distress score ranging from 0-42, and two subscales consisting of seven items each: anxiety (range 0-21) and depression (range 0-21). Higher scores reflect greater distress. The HADS will be administered with a set of questionnaires in the first hour of the two-hour session.
Buckley Scale (baseline) | In the first hour of the two-hour session
  The Buckley Scale is a 12-item measure designed to assess feelings of happiness, anxiety, anger, sadness, and hurt feelings in the present moment. The scale is composed of five subscales for these five domains of emotion. Respondents indicate the degree to which they endorse a particular feeling using a seven-point Likert scale ranging from "not at all" to "extremely," with higher scores reflecting more intensity of each of the aforementioned emotions. The Buckley Scale will be administered with a set of questionnaires in the first hour of the two-hour session.
Buckley Scale (change) | Within the first hour and again within the final 30 minutes of the two-hour session.
  The Buckley Scale is a 12-item measure designed to assess feelings of happiness, anxiety, anger, sadness, and hurt feelings in the present moment. The scale is composed of five subscales for these five domains of emotion. Respondents indicate the degree to which they endorse a particular feeling using a seven-point Likert scale ranging from "not at all" to "extremely," with higher scores reflecting more intensity of each of the aforementioned emotions. Change in Buckley Scale will be calculated by determining the difference between Buckley Scale score at baseline and score from when it is administered again within the final 30 minutes of the two-hour session.
Binge Eating Scale | In the first hour of the two-hour session
  The Binge Eating Scale (BES) is a 16-item questionnaire designed to assess the behavioral (e.g., large amount of food consumed), as well as the cognitive and emotional (e.g., feeling out of control while eating), features of binge eating. Respondents select one of three or four response options coded 0 to 2 or 3, respectively. Scores are summed and range from 0 to 46, with higher scores reflecting more severe binge eating problems. The BES will be administered with a set of questionnaires in the first hour of the two-hour session.
Vividness of Recall | Immediately following weight stigma vignette in the final 30 minutes of the two-hour session.
  A single-item measure will be administered to assess vividness of participants' recall of the instance when they themselves experienced weight stigmatization that they write about in the weight stigma induction.

CONTACTS AND LOCATIONS:
Overall Officials: Charles F Emery, Ph.D., Principal Investigator — Professor and Psychology Department Chair
Locations (1):
- The Ohio State University, Columbus, Ohio, United States

IPD SHARING:
Plan to Share IPD: Undecided

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-11-24): https://cdn.clinicaltrials.gov/large-docs/26/NCT04573426/Prot_SAP_000.pdf